CLINICAL TRIAL: NCT05425758
Title: What is the Optimal Index for Assessment of Plaster Cast Quality in Pediatric Distal Forearm Fractures
Brief Title: Optimal Index for Pediatric Distal Forearm Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Meena Mikhael Rizk, Principal Investigator of orthopedic surgery, Sohag University
Other Study IDs: Soh-Med-22-05-07
Record Dates: First submitted 2022-06-11; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pediatric Distal Forearm Fractures
Keywords: Optimal index for Pediatric distal forearm fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective radiographic study of displaced distal forearm fractures requiring manipulation for children 3-12 years of age and will be treated with casting.The patients' full radiographic series (including the pre-manipulation, immediate post-manipulation, after 1 week and after 4 weeks radiographs) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 3 to 12 years old.
2. Any presentation of displaced distal forearm fractures requiring manipulation and will be treated with casting.

Exclusion Criteria:

1. Children with compound fractures (those with unacceptable initial reduction, fracture dislocations, and fractures with physeal separation) will be excluded from the study, as those will be treated with Kirschner wires.
2. Children whose casts is split will be excluded.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 3-12 years of age with displaced distal forearm fractures requiring manipulation for and will be treated with casting.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The cast index | 4 weeks observation after reduction and applying cast.
  formula that use measurements obtained from anteroposterior and lateral plain radiographs to estimate the quality of cast placement.
The gap index | 4 weeks observation after reduction and applying cast.
  formula that use measurements obtained from anteroposterior and lateral plain radiographs to estimate the quality of cast placement.
The padding index | 4 weeks observation after reduction and applying cast.
  formula that use measurements obtained from anteroposterior and lateral plain radiographs to estimate the quality of cast placement.
The Canterbury index | 4 weeks observation after reduction and applying cast.
  formula that use measurements obtained from anteroposterior and lateral plain radiographs to estimate the quality of cast placement.
The three-point index | 4 weeks observation after reduction and applying cast.

IPD SHARING:
Plan to Share IPD: Undecided